CLINICAL TRIAL: NCT03755141
Title: Open Label, Multicenter, Prospective Phase II Study to Investigate the Efficacy and Safety of Trastuzumab Biosimilar (Herzuma®) Plus Treatment of Physician's Choice (TPC) in Patients With HER-2 Positive Metastatic Breast Cancer Who Progressed After 2 or More HER-2 Directed Chemotherapy
Brief Title: Efficacy and Safety of Trastuzumab Biosimilar (Herzuma®) Plus Treatment of Physician's Choice (TPC) in Patients With HER-2 Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, In Hae Park, Senior Scientist, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM10B
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Herzuma (Experimental): Herzuma + TPC
  Interventions: Drug: Herzuma

INTERVENTIONS:
Drug: Herzuma — Herzuma + Treatment of Physician's Choice

SUMMARY:
Trastuzumab combined with chemotherapy has been approved as the first line therapy in HER2+ metastatic breast cancer. When patients experienced progression beyond trastuzumab containing therapy, T-DM1 is considered as the second line therapy followed by trastuzumab plus any other chemotherapeutic agents or lapatinib plus capecitabine.

A biosimilar drug is a biological product that is highly similar to a licensed biological product, with no clinically meaningful differences in terms of safety, purity, or potency. Several trastuzumab biosimilar products have been approved after efficacy and safety studies which were usually as the first line setting with taxane combined.

Even though trastuzumab biosimilar drugs demonstrated similarity of equivalence with trastuzumab in these studies, the efficacy of their second use beyond progression with other chemotherapeutic agents has not been tested yet. In addition, the investigators don't have any data regarding possible cross reactivity between trastuzumab and trastuzumab biosimilar drugs.

In this study, the investigators plan multicenter phase II clinical trial to test the efficacy, safety and immunogenicity of trastuzumab biosimilar, Herzuma® in combination with TPC in patients with HER2+ metastatic breast cancer who progressed after 2 or more HER-2 directed chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult, ≥ 19 years old at the time of informed consent.
2. Patient has histologically and/or cytologically confirmed diagnosis of HER2-positive breast cancer (HER-2/neu 3+ as defined by immunohistochemistry and/or HER-2/neu gene amplification as defined by fluorescence in situ hybridization).
3. Metastatic or unresectable disease documented on diagnostic imaging studies.
4. Prior 2 or more HER-2 directed therapy for metastatic disease is mandatory.
5. Patient must have at least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
7. Adequate bone marrow and organ function including: a) WBC ≥ 3500/ml; b) Platelets ≥ 100,000/ul; c) Hemoglobin >9.0 g/dl; d) Total bilirubin ≤ 1.5x ULN; e) AST and ALT < 2.5 x ULN; f) Alkaline phosphatase <2.5x ULN; g) Creatinine ≤ 1.5x ULN or CCr >60 ml/min for patients with abnormal serum Cr level function.
8. Life expectance longer than 3 months
9. Patient has an adequate left ventricular ejection function of at least 55 % at baseline, as measured by echocardiography.
10. Written informed consent

Exclusion Criteria:

1. Patient is pregnant or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
2. Patient has symptomatic and unstable CNS metastases, except for treated brain metastases. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed.
3. Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus syndrome (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness. Baseline viral assessment is not required in patients with no known infection.
4. Major surgery within 4 weeks of first dose of investigational product or not fully recovered from any side effects of previous procedures.
5. Any other malignancy within 3 years prior to first dose of investigational product except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
6. QTc interval >480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.
7. Any of the following within 6 months of first dose of investigational product myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE v. 5.0 Grade ≤2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
8. History of symptomatic interstitial pneumonitis.
9. Patients with a history of hypersensitivity reactions to trastuzumab, rodent-derived proteins, or components of trastuzumab.
10. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In Hae Park, MD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University, Guro hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
safety profiles, efficacy data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Herzuma
Started | 109 (A total of 109 patients were enrolled during study period .)
Completed | 109 (A total of 109 patients were enrolled in Herzuma arm.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: HER2+ metastatic breast cancer
Arm/Group | Herzuma
Number analyzed (Participants) | 109
Age, Continuous [Median (Full Range); unit: years] | 55 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 109
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 109

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: defined as the time from study entry until the first observation of existing disease progression according to the above schedule or death due to any cause.
Time Frame: 6 months after last patient enrollment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Herzuma
Number analyzed (Participants) | 109
months | 4.6 [2.8 to 7.2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Herzuma
All-Cause Mortality (participants affected / at risk) | 37/109
Serious Adverse Events (participants affected / at risk) | 42/109
Other Adverse Events (participants affected / at risk) | 29/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herzuma (N=109)
cardiac event (Cardiac disorders) | 1
hematologic event (Blood and lymphatic system disorders) | 39
non-hematologic event (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herzuma (N=109)
hematologic event (Blood and lymphatic system disorders) | 17
non-hematologic event (Gastrointestinal disorders) | 10
cardiac event (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03755141/Prot_SAP_000.pdf